CLINICAL TRIAL: NCT00924703
Title: Long-term Extension of a Phase 2, Open-Label Dose-Finding Study to Evaluate the Safety, Efficacy, and Tolerability of Multiple Subcutaneous Doses of rAvPAL-PEG in Subjects With PKU
Brief Title: Long-Term Extension of Previous rAvPAL-PEG Protocols in Subjects With PKU (PAL-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-003
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Phenylketonuria
MeSH Terms: conditions — Phenylketonurias | interventions — pegvaliase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rAvPAL-PEG (Experimental): rAvPAL-PEG in varying doses dependent on safety and efficacy.
  Interventions: Drug: rAvPAL-PEG

INTERVENTIONS:
Drug: rAvPAL-PEG — The doses are planned to be in the same range as those tested in PAL-002 or PAL-004 and then modified either by increasing or decreasing the dose, adhering to an upper limit up to 5.0 mg/kg per week or 375 mg/week, considering each subject's individual responses related to safety and efficacy.
  Other Names: Pegvaliase

SUMMARY:
This study is an extension of previous rAvPAL-PEG studies. Administration of rAvPAL-PEG will be continued to assess whether long-term dosing of rAvPAL-PEG is safe and can maintain reduced blood Phe concentrations in PKU subjects.

DETAILED DESCRIPTION:
PAL-003 is designed to evaluate long-term treatment of subjects who are continuing to take rAvPAL-PEG. Subjects'previous rAvPAL-PEG dosing will continue in PAL-003. In PAL-003, each subject's dose will be adjusted as needed to attain or maintain blood Phe concentrations of 60-600 µmol/L. rAvPAL-PEG dose will be based on either a subject's weight or will be a fixed dose (subjects who have maintained blood Phe levels to 60-600 µmol/L for at least 2 consecutive weeks and who have maintained a stable rAvPAL-PEG dose for at least 2 consecutive weeks). Doses will be evaluated on an individual basis.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed participation in previous rAvPAL-PEG studies.
* Willing and able to provide written, signed informed consent, or, in the case of participants under the age of 18, provide written assent (if required) and written informed consent by a parent or legal guardian, after the nature of the study has been explained, and prior to any research-related procedures.
* Willing and able to comply with all study procedures.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have been in menopause at least 2 years, or had tubal ligation at least 1 year prior to Screening, or who have had total hysterectomy.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Maintained a stable diet.
* In generally good health as evidenced by physical examination, clinical laboratory evaluations (hematology, chemistry, and urinalysis), and electrocardiogram (ECG) at Screening.

Exclusion Criteria:

* Use of any investigational product (with the exception of rAvPAL-PEG) or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Use of any medication that is intended to treat PKU within 14 days prior to the administration of study drug.
* Use or planned use of any injectable drugs containing PEG (other than rAvPAL-PEG), including Depo-Provera during study participation.
* A prior reaction that included systemic symptoms (eg, generalized hives, respiratory or gastrointestinal problems, hypotension, angioedema, anaphylaxis) to rAvPAL-PEG or a PEG-containing product.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) or to breastfeed at any time during the study.Concurrent disease or condition that would interfere with study participation or safety (eg, history or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurological, oncologic, or psychiatric disease).
* Any condition that, in the view of the PI, places the subject at high risk of poor treatment compliance or of not completing the study.
* Known hypersensitivity to rAvPAL-PEG or its excipients, including hypersensitivity reactions that necessitated early termination from previous rAvPAL-PEG studies.
* Alanine aminotransferase (ALT) concentration > 2 times the upper limit of normal.
* Creatinine > 1.5 times the upper limit of normal.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2010-01-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (14):
- United States (14):
  - The Children's Hospital, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - Ann and Robert H Lurie Children's Hospital, Chicago, Illinois
  - University of Louisville, Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Washington University Center for Applied Research Sciences, St Louis, Missouri
  - Nebraska Medical Center, Omaha, Nebraska
  - Albany Medical Center, Albany, New York
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Utah Hospital, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burton BK, Longo N, Vockley J, Grange DK, Harding CO, Decker C, Li M, Lau K, Rosen O, Larimore K, Thomas J; PAL-002 and PAL-004 Investigators. Pegvaliase for the treatment of phenylketonuria: Results of the phase 2 dose-finding studies with long-term follow-up. Mol Genet Metab. 2020 Aug;130(4):239-246. doi: 10.1016/j.ymgme.2020.06.006. Epub 2020 Jun 16. PMID 32593547
- [Derived] Longo N, Zori R, Wasserstein MP, Vockley J, Burton BK, Decker C, Li M, Lau K, Jiang J, Larimore K, Thomas JA. Long-term safety and efficacy of pegvaliase for the treatment of phenylketonuria in adults: combined phase 2 outcomes through PAL-003 extension study. Orphanet J Rare Dis. 2018 Jul 4;13(1):108. doi: 10.1186/s13023-018-0858-7. PMID 29973227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study, conducted in 14 study centers of United States.
Groups:
- rAvPAL-PEG: rAvPAL-PEG 0.001 to a maximum dose of 5.0 mg/kg/week or 375 mg/week by subcutaneous injection
Period: Overall Study
Arm/Group | rAvPAL-PEG
Started | 68
Completed | 46
Not Completed | 22
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 5
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Sponsor | 1

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.31 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  White | 66
  Asian | 1
Weight [Mean (Standard Deviation); unit: kg] | 83.0 (26.39)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Total 5 (7.4%) out of 68 subjects BMI are missing due to missing height
  kg/m^2
    number analyzed (Participants) | 63
    (all) | 29.2 (8.44)
Baseline blood Phe [Mean (Standard Deviation); unit: μmol/L] | 1022.4 (530.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Blood Phenylalanine (Phe) Concentration
Description: Blood Phe Concentration (Change from Baseline) and Daily Dose in PAL-003 Subjects by Disposition (PAL-003 Population)
Time Frame: At Baseline and Change from Baseline to Week 48, Week 96, Week 144, Week 216, and Week 240
Population: Efficacy population consisted of all subjects who received at least one dose of study drug and have post-treatment blood Phe concentration measurements.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 68
μmol/L
  Baseline | 1022.4 (530.39)
  Change from Baseline to Week 48: number analyzed (Participants) | 60
  Change from Baseline to Week 48 | -553.5 (652.95)
  Change from Baseline to Week 96: number analyzed (Participants) | 53
  Change from Baseline to Week 96 | -653.3 (637.81)
  Change from Baseline to Week 144: number analyzed (Participants) | 44
  Change from Baseline to Week 144 | -672.3 (621.06)
  Change from Baseline to Week 216: number analyzed (Participants) | 31
  Change from Baseline to Week 216 | -535.9 (573.08)
  Change from Baseline to Week 240: number analyzed (Participants) | 29
  Change from Baseline to Week 240 | -574.9 (549.90)

2. Secondary Outcome: Pharmacokinetics-Plasma Pegvaliase Concentration
Description: Steady-state Pharmacokinetics (PK) of pegvaliase was measured in subjects who have achieved and maintained target blood Phe
Time Frame: At Baseline, Week 48, Week 96, Week 144, Week 216 and Week 240
Population: As PAL-003 is an extension of parent Phase 2 studies (PAL-002, PAL-004 & 165-205), the parent Phase 2 treatment naïve baseline data (N=80) was used for the vital signs, immunogenicity & PK analyses to monitor changes in vital signs mediated by pegvaliase, understand development & maturation of immune response against pegvaliase, & the resulting impact on PK. Refer to NCT00925054-PAL-002, NCT01212744-PAL-004 & NCT01560286-165-205 for parent Ph2 demographic data (N=80).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 80
ng/mL
  At Baseline: number analyzed (Participants) | 39
  At Baseline | 961.5 (3013.43)
  Week 48: number analyzed (Participants) | 53
  Week 48 | 4127.3 (6116.72)
  Week 96: number analyzed (Participants) | 44
  Week 96 | 7457.7 (10685.02)
  Week 144: number analyzed (Participants) | 45
  Week 144 | 7196.1 (11678.89)
  Week 216: number analyzed (Participants) | 28
  Week 216 | 7764.4 (9292.34)
  Week 240: number analyzed (Participants) | 29
  Week 240 | 6557.8 (9220.95)

3. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: A treatment-emergent AE was defined as any adverse event (AE) newly appearing or worsened in severity following initiation of study drug until 4 weeks after last dose of pegvaliase (PAL-003)
Time Frame: Up to 109 months.
Population: Analysis population consisted of subjects from the study of PAL-003 only
Measure: Count of Participants; unit: Participants
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 68
Participants
  Subjects with any adverse event | 68
  Subjects with any serious adverse events | 12
  Subjects with any treatment-related adverse event | 65
  Any treatment-related serious adverse event | 6
  Death | 0

4. Secondary Outcome: Percentage of Participants With Positive PEG IgG Antibody
Description: The presence of IgG Antibodies against PEG (polyethylene glycol) is measured overtime
Time Frame: At Baseline and Change from Baseline to Week 24, Week 52, Week 104 and Week 156
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 80
Participants
  Baseline: number analyzed (Participants) | 79
  Baseline | 29
  Change from Baseline to Week 24: number analyzed (Participants) | 64
  Change from Baseline to Week 24 | 24
  Change from Baseline to Week 52: number analyzed (Participants) | 60
  Change from Baseline to Week 52 | 14
  Change from Baseline to Week 104: number analyzed (Participants) | 48
  Change from Baseline to Week 104 | 2
  Change from Baseline to Week 156: number analyzed (Participants) | 45
  Change from Baseline to Week 156 | 7

5. Secondary Outcome: Percentage of Participants With Positive PAL IgG Antibody
Description: The presence of IgG Antibodies against PAL (phenylalanine ammonia lyase) is measured overtime
Time Frame: At Baseline and Change from Baseline to Week 24, Week 52, Week 104 and Week 156
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | rAvPAL-PEG
Number analyzed (Participants) | 80
Participants
  Baseline: number analyzed (Participants) | 79
  Baseline | 10
  Change from Baseline to Week 24: number analyzed (Participants) | 64
  Change from Baseline to Week 24 | 63
  Change from Baseline to Week 52: number analyzed (Participants) | 60
  Change from Baseline to Week 52 | 60
  Change from Baseline to Week 104: number analyzed (Participants) | 48
  Change from Baseline to Week 104 | 48
  Change from Baseline to Week 156: number analyzed (Participants) | 45
  Change from Baseline to Week 156 | 45

ADVERSE EVENTS:
Time Frame: Up to 109 months.
Description: Only treatment-emergent AEs that occurred and were reported during the study period were included in AE summaries. The incidence, exposure-adjusted event rate, severity grade (assessed per CTCAE version 4.03), and relationship to study drug (per Investigator) for all treatment-emergent AEs were summarized. For AEs occurring more than once during the study, maximum severity was used to summarize AEs by severity.
Arm/Group | rAvPAL-PEG
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 12/68
Other Adverse Events (participants affected / at risk) | 68/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAvPAL-PEG (N=68)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAvPAL-PEG (N=68)
Lymphadenopathy (Blood and lymphatic system disorders) | 9 (12)
Injection site reaction (General disorders) | 36 (114)
Injection site erythema (General disorders) | 36 (160)
Injection site bruising (General disorders) | 34 (245)
Pyrexia (General disorders) | 25 (38)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 25 (59)
Injection site rash (General disorders) | 11 (24)
Injection site pruritus (General disorders) | 22 (83)
Injection site pain (General disorders) | 18 (76)
Injection site swelling (General disorders) | 16 (25)
Injection site urticaria (General disorders) | 18 (66)
Fatigue (General disorders) | 17 (24)
Peripheral swelling (General disorders) | 9 (18)
Pain (General disorders) | 15 (22)
Toothache (Gastrointestinal disorders) | 13 (20)
Fall (Injury, poisoning and procedural complications) | 7 (7)
Procedural pain (Injury, poisoning and procedural complications) | 7 (10)
Injection site mass (General disorders) | 5 (9)
Injection site nodule (General disorders) | 5 (8)
Injection site discolouration (General disorders) | 4 (17)
Injection site haemorrhage (General disorders) | 4 (6)
Headache (Nervous system disorders) | 43 (253)
Dizziness (Nervous system disorders) | 26 (61)
Contusion (Injury, poisoning and procedural complications) | 24 (59)
Anxiety (Psychiatric disorders) | 12 (17)
Migraine (Nervous system disorders) | 14 (41)
Hypertension (Vascular disorders) | 9 (9)
Oedema peripheral (General disorders) | 4 (10)
Vertigo (Ear and labyrinth disorders) | 4 (5)
Insomnia (Psychiatric disorders) | 14 (30)
Depression (Psychiatric disorders) | 13 (16)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (11)
Irritability (Psychiatric disorders) | 6 (9)
Disturbance in attention (Nervous system disorders) | 5 (5)
Rash generalised (Skin and subcutaneous tissue disorders) | 6 (17)
Arthropod bite (Injury, poisoning and procedural complications) | 11 (14)
Paraesthesia (Nervous system disorders) | 8 (12)
Seasonal allergy (Immune system disorders) | 5 (9)
Influenza like illness (General disorders) | 6 (10)
Tendonitis (Musculoskeletal and connective tissue disorders) | 4 (7)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 11 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (12)
Thermal burn (Injury, poisoning and procedural complications) | 9 (11)
Skin abrasion (Injury, poisoning and procedural complications) | 7 (9)
Acne (Skin and subcutaneous tissue disorders) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Rash (Skin and subcutaneous tissue disorders) | 38 (124)
Urticaria (Skin and subcutaneous tissue disorders) | 33 (294)
Pruritus (Skin and subcutaneous tissue disorders) | 27 (69)
Erythema (Skin and subcutaneous tissue disorders) | 14 (31)
Rash erythematous (Skin and subcutaneous tissue disorders) | 16 (21)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (14)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (6)
Nasopharyngitis (Infections and infestations) | 45 (137)
Upper respiratory tract infection (Infections and infestations) | 34 (157)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 22 (43)
Urinary tract infection (Infections and infestations) | 14 (21)
Gastroenteritis viral (Infections and infestations) | 12 (21)
Influenza (Infections and infestations) | 13 (18)
Pharyngitis streptococcal (Infections and infestations) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Viral infection (Infections and infestations) | 8 (14)
Gastroenteritis (Infections and infestations) | 7 (16)
Asthenia (General disorders) | 4 (5)
Fungal infection (Infections and infestations) | 4 (7)
Nephrolithiasis (Renal and urinary disorders) | 6 (7)
Microalbuminuria (Renal and urinary disorders) | 4 (8)
Proteinuria (Renal and urinary disorders) | 4 (4)
Alanine aminotransferase increased (Investigations) | 4 (7)
Amino acid level decreased (Investigations) | 4 (5)
Ear infection (Infections and infestations) | 5 (6)
Ear pain (Ear and labyrinth disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (52)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 33 (82)
Sinusitis (Infections and infestations) | 25 (41)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 15 (33)
Chest discomfort (General disorders) | 8 (12)
Laceration (Injury, poisoning and procedural complications) | 10 (18)
Bronchitis (Infections and infestations) | 9 (12)
Chest pain (General disorders) | 5 (6)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Raynaud's phenomenon (Vascular disorders) | 5 (6)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Complement factor C3 decreased (Investigations) | 7 (8)
Dysmenorrhoea (Reproductive system and breast disorders) | 9 (42)
Complement factor C4 decreased (Investigations) | 7 (9)
Hypoaesthesia (Nervous system disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Blood uric acid increased (Investigations) | 5 (6)
Haematuria (Renal and urinary disorders) | 6 (8)
Amino acid level increased (Investigations) | 5 (5)
Blood bicarbonate decreased (Investigations) | 4 (4)
Urobilinogen urine increased (Investigations) | 4 (4)
Eye swelling (Eye disorders) | 5 (7)
Ocular hyperaemia (Eye disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 33 (70)
Vomiting (Gastrointestinal disorders) | 30 (64)
Diarrhoea (Gastrointestinal disorders) | 27 (79)
Abdominal pain (Gastrointestinal disorders) | 20 (42)
Abdominal pain upper (Gastrointestinal disorders) | 13 (31)
Dyspepsia (Gastrointestinal disorders) | 11 (21)
Abdominal discomfort (Gastrointestinal disorders) | 13 (26)
Constipation (Gastrointestinal disorders) | 8 (10)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (7)
Food poisoning (Gastrointestinal disorders) | 5 (8)
Dental caries (Gastrointestinal disorders) | 5 (6)
Tooth abscess (Infections and infestations) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 (188)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (78)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (67)
Neck pain (Musculoskeletal and connective tissue disorders) | 18 (27)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 (28)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 13 (20)
Joint swelling (Musculoskeletal and connective tissue disorders) | 10 (12)
Ligament sprain (Injury, poisoning and procedural complications) | 10 (12)
Tremor (Nervous system disorders) | 5 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (12)
Non-cardiac chest pain (General disorders) | 4 (4)
Joint dislocation (Injury, poisoning and procedural complications) | 4 (4)
Wound (Injury, poisoning and procedural complications) | 4 (6)
Folliculitis (Infections and infestations) | 4 (6)
Vessel puncture site bruise (General disorders) | 4 (9)
Muscle strain (Injury, poisoning and procedural complications) | 5 (5)
Injection site induration (General disorders) | 4 (9)
Abdominal distension (Gastrointestinal disorders) | 4 (9)
Adverse drug reaction (General disorders) | 5 (10)
Hypersensitivity (Immune system disorders) | 4 (5)
Joint injury (Injury, poisoning and procedural complications) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT00924703/Prot_000.pdf
  • Statistical Analysis Plan (2016-04-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT00924703/SAP_001.pdf